CLINICAL TRIAL: NCT02408731
Title: A Randomized, Double-blind, Placebo-controlled Phase I Study to Determine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of PMZ-2010 (Centhaquin) in Healthy Male Volunteers
Brief Title: A Study to Determine the Safety, Tolerability and Pharmacokinetics of PMZ-2010 (Centhaquin) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-430-CENT-2012
Record Dates: First submitted 2015-03-20; First posted 2015-04-03 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
MeSH Terms: interventions — centhaquine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Single dose of 0.005 mg/kg of PMZ-2010 (Experimental): A single dose of 0.005 mg/kg of PMZ-2010 (n=3) or placebo (n=1)
  Interventions: Drug: PMZ-2010 (Centhaquin)
- Single dose of 0.01 mg/kg of PMZ-2010 (Experimental): A single dose of 0.01 mg/kg of PMZ-2010 (n=3) or placebo (n=1)
  Interventions: Drug: PMZ-2010 (Centhaquin)
- Single dose of 0.05 mg/kg of PMZ-2010 (Experimental): A single dose of 0.05 mg/kg of PMZ-2010 (n=3) or placebo (n=1)
  Interventions: Drug: PMZ-2010 (Centhaquin)
- Single dose of 0.10 mg/kg of PMZ-2010 (Experimental): A single dose of 0.10 mg/kg of PMZ-2010 (n=3) or placebo (n=1)
  Interventions: Drug: PMZ-2010 (Centhaquin)
- 3 doses equivalent to MTD of PMZ-2010 (Experimental): Three equally divided doses (total dose/day equivalent to MTD) of PMZ-2010 (n=3) or placebo (n=1) for 2 days
  Interventions: Drug: PMZ-2010 (Centhaquin)
- 3 doses equivalent to 2*MTD of PMZ-2010 (Experimental): Three equally divided doses (total dose/day equivalent to 2*MTD) of PMZ-2010 (n=3) or placebo (n=1) for 2 days
  Interventions: Drug: PMZ-2010 (Centhaquin)

INTERVENTIONS:
Drug: PMZ-2010 (Centhaquin) — As per the randomization schedule, injection of PMZ-2010 or placebo (100 ml normal saline) will be administered to each subject under supervision of investigator as an intravenous infusion over one hour. PMZ-2010 will be dissolved in normal saline (100 ml) before administration.
  Other Names: Placebo (normal saline)

SUMMARY:
Shock is a condition of reduced tissue perfusion, resulting in the inadequate delivery of oxygen and nutrients that are necessary for cellular function. The current resuscitative agents can extend patient's life to a limited extent. Centhaquin (PMZ-2010) in very low doses reduced blood lactate levels, improved blood pressure, cardiac output, survival and proved to be a highly effective resuscitative agent. The investigators are conducting a phase I clinical study in humans to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of centhaquin citrate in normal healthy volunteers.

DETAILED DESCRIPTION:
Shock is a condition of reduced tissue perfusion, resulting in the inadequate delivery of oxygen and nutrients that are necessary for cellular function. Common causes of shock are hypovolemia (excessive blood or fluid loss), sepsis, cardiac failure, dengue and neuroendocrine dysfunction. The current resuscitative measures include administration of crystalloid solutions (e.g., 0.9% saline, Ringer's lactate, or hypertonic saline) or colloid solutions (e.g., hydroxyethyl starch, albumin, or dextrans). These agents can extend patient's life to a limited extent. Centhaquin (PMZ-2010) in very low doses reduced blood lactate levels, improved blood pressure, cardiac output, survival and proved to be a highly effective resuscitative agent. The investigators are conducting a phase I clinical study in humans to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of centhaquin citrate in normal healthy volunteers. Successful completion of phase I studies will lead to efficacy studies in patients with hypovolemic shock.

ELIGIBILITY:
Inclusion Criteria: Subjects to be enrolled in this trial must fulfill all of these criteria:

* Sex: male
* Age: 18-60 yr old, both inclusive
* Having a Body Mass Index (BMI) between 18.5-28 kg / m2 (both inclusive) and body weight not less than 45 kg
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; and to comply with the requirements of the entire study
* Voluntarily given written informed consent to participate in this study
* Be of normal health as determined by the principal investigator from medical history, physical examination and laboratory investigations, 12-lead ECG and X-ray chest of the subjects performed within 10 days prior to the admission of the study
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, coke, chocolate, "power drinks") and grapefruit (juice) from 48 h prior to each admission until study completion

Exclusion Criteria: Subjects meeting any of these criteria will not be enrolled in the study:

* Employees of JCDC or Pharmazz India Private Limited
* Not willing to use contraceptives (preferably condoms) during sexual activity for the period of 3 months from the date of check-in
* History of hypersensitivity and / or intolerance to Centhaquin or any other related compounds.
* History of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study.
* Clinically abnormal ECG and Chest X-ray.
* Physical findings: clinically relevant abnormal physical findings (including body temperature) suggesting underlying pathologies or those which could interfere with the objectives of the study.
* Subjects with impaired renal function as measured by glomerular filtration rate <90 mL/min/1.73m2 estimated using the modification of diet in renal disease (MDRD) formula [GFR for Male =186 × (Serum Creatinine)-1.154 × Age-0.203 ]12
* Laboratory values that are significantly different than the normal reference range and/or are deemed to be of clinical significance by the investigator
* Presence of reactive disease markers of HIV 1 and II, HBsAg, HCV or VDRL.
* Positive for alcohol breath test and/or urine drug screen (barbiturates, benzodiazepines, amphetamine, cocaine, opiates, tetra-hydro cannabinol).
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Diseases: relevant history of renal, hepatic, cardiovascular, respiratory, skin, haematological, endocrine, neurological or gastrointestinal diseases. History of depression, psychosis, schizophrenia or any other severe psychiatric diseases, or epilepsy, or any other illness that may interfere with the aim of the study. History of any significant illness in the 4 weeks preceding the screening
* Medications: history of intake of any medications including over the counter medications (OTC) and any herbal agents at least 4 weeks period prior to study drug administration.
* Investigational drug trials: participation in the evaluation of any drug in the 3 months prior to the start of the study (dosing with IMP).
* Blood donation: Subjects who, through completion of this study, would have donated and/or lost more than 300 mL of blood in the past 12 weeks Note: In case the blood loss is ≤ 200 mL; subject may be dosed 60 days after blood donation or last sample of the previous study
* Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or alcoholics

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 7 days
  Measure blood pressure, heart rate, body temperature, ECG, laboratory parameters and clinical assessment.after single and multiple ascending doses of PMZ-2010.

SECONDARY OUTCOMES:
Composite of pharmacokinetics of PMZ-2010 in plasma | 24 hours
  Maximum concentration (Cmax), Time of maximum plasma concentration (Tmax), Area under the concentration-time curve (AUC) from time of dosing to the last quantifiable concentration (AUClast), Terminal elimination half-life (t½), Clearance (CL/F), Apparent volume of distribution during the terminal elimination phase (Vz/F) of PMZ-2010 in plasma after single ascending doses.
Phamacodynamics profile of PMZ-2010 | 7 days
  Change in systolic and diastolic blood pressure, pulse rate, heart rate, QTcF after single ascending dose and multiple ascending doses

CONTACTS AND LOCATIONS:
Overall Officials: Ashish O Goyal, MD, Principal Investigator — Jehangir Clinical Development Centre Pvt. Ltd.
Locations (1):
- Jahangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra, India

REFERENCES:
- [Background] Gulati A, Zhang Z, Murphy A, Lavhale MS. Efficacy of centhaquin as a small volume resuscitative agent in severely hemorrhaged rats. Am J Emerg Med. 2013 Sep;31(9):1315-21. doi: 10.1016/j.ajem.2013.05.032. Epub 2013 Jul 19. PMID 23871440
- [Background] Lavhale MS, Havalad S, Gulati A. Resuscitative effect of centhaquin after hemorrhagic shock in rats. J Surg Res. 2013 Jan;179(1):115-24. doi: 10.1016/j.jss.2012.08.042. Epub 2012 Sep 2. PMID 22964270
- [Background] Gulati A, Lavhale MS, Garcia DJ, Havalad S. Centhaquin improves resuscitative effect of hypertonic saline in hemorrhaged rats. J Surg Res. 2012 Nov;178(1):415-23. doi: 10.1016/j.jss.2012.02.005. Epub 2012 Apr 2. PMID 22487389